CLINICAL TRIAL: NCT03072004
Title: Evaluation of Low Level Laser Therapy Effects in Peripheral Nerves Patient Affected With Leprosy : Randomized Controlled Trial
Brief Title: Low Level Laser Therapy Effects in Peripheral Nerves Patient With Leprosy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Elaine Fávaro Pípi Sabino, Principal Investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 37474214.4.0000.5152
Record Dates: First submitted 2017-02-14; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Leprosy Neuropathy
Keywords: Leprosy; Neuropathy; LLLT
MeSH Terms: conditions — Leprosy | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: We will analyze leprosy patients with neuropathy. These patients will be randomly divided in: (a) Control: who will receive simulated application "sham" of LLLT; and (b) LLLT: who will receive LLLT (830 nm, continuous emission, 100mW output power and 3J power density). Treatments will occur in 12 sessions (3 times per week) on the nerves: a)ulnar: around the ulnar nerve at the elbow region, and b)common peroneal: surrounding fibular head. For the inclusion criteria will be selected leprosy patients (tuberculoid and borderline tuberculoid forms) with focal demyelinating neuropathy of the ulnar and common peroneal nerves by electroneuromyography (ENMG); patients without leprosy reactions and corticoid use. We will perform measurements of the following parameters before and after the LLLT protocol application: ENMG Muscle Strength; Tactile Sensitivity measured; Pain Intensity; Incapacity grade; Infrared thermography; Screening of Activity Limitation and Safety Awareness scale.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Leprosy patients with focal demyelinating neuropathy in compression sites of the ulnar and common peroneal nerves who will receive application "sham LLLT". The laser will be turned off, but the procedure will be the same as with the Low Level Laser Therapy (LLLT) group
  Interventions: Device: Sham LLLT
- Low Level Laser Therapy (Experimental): Leprosy patients with focal demyelinating neuropathy in compression sites of the ulnar and common peroneal nerves who will receive intervention with low-intensity laser therapy (LLLT).
  Interventions: Device: LLLT

INTERVENTIONS:
Device: LLLT — The LLLT will be applied using a diode laser device (Recover Laser MMOptics, São Carlos/SP- Brazil) with parameters: 808nm, continuous output, 100mW, 8J. Laser probe will be applied directly and perpendicularly in skin contact (5 points), the time of irradiation will be 80 seconds per point, and treatments will be applied for three times a week for 12 sessions.
  Arms: Low Level Laser Therapy
Device: Sham LLLT — That group receive application "sham LLLT". The laser will be turned off, but the procedure will be the same as with the LLLT group
  Arms: Control

SUMMARY:
We are going to investigate leprosy patients with neuropathies. This problem can lead to changes in nerve function and lead to disability. We will investigate a protocol with LLLT to improve pain, inflammation, and to prevent disabilities. We will test two groups, which will be divided into control and LLLT treated patients. In this groups we will perform quantitative measurements of the following parameters before and after the protocol application: electroneuromyography and muscle strength measurements, evaluation of activity limitation and risk awareness, evaluation of tactile sensitivity and evaluation of temperatures of hands and feet. Averages for all parameters will be compared before and after treatment (12 application sessions). We believe that LLLT can become an important alternative treatment to improve conduction velocity, tactile sensitivity, temperatures of hands and feet, muscle strength and pain, which will prevent nerve damage and disabilities

DETAILED DESCRIPTION:
Leprosy is an infectious disease caused by Mycobacterium leprae, which is an obligate intracellular bacillus with the capacity to invade cells of the peripheral nervous system (Nations et al., 1998). This disease presents polymorphic clinical features, and the destruction of peripheral nerves is relevant, resulting in irreversible disabilities with great social and psychological impact (Martins et al., 2008).

Among the 250,000 new cases of leprosy detected worldwide every year, 12% to 55% demonstrate diagnosis of sensory, motor or autonomic neuropathy (Saunderson et al., 2000). The destruction of nerve fibers in patients with leprosy can be established by the presence of inflammatory process and the development of autoimmunity and cytotoxicity (Birdi et al., 1996), including nerve growth factor (Facer et al., 1998), glia cells' adhesion molecules, interferon-gamma,Transforming Growth Factor - Beta (Goulart et al., 1996; Goulart et al., 2000), Tumor Necroses Factor-alpha (Singh, 1998) and interleukins (IL-6, IL-8, IL-12 and IL-10) (Mendonça et al., 2008).

Low Level Laser Therapy (LLLT) has been demonstrated as a promising treatment in neural rehabilitation. Some studies, has demonstrated that LLLT presented positive results in improving nerve conduction velocity. The literature has provided evidences for the effectiveness of LLLT treatment in neural rehabilitation, and it may be a promising tool for leprosy neuropathies rehabilitation.

LLLT provided improvements in clinical and electrophysiological parameters in humans with ulnar neuropathy and this modality showed a satisfying short-term effectiveness in the treatment of this pathology (Ozkan et al., 2014). Other studies have shown that the LLLT application in diabetic polyneuropathy presented positive results in improving nerve conduction velocity (Khamseh et al., 2011).

Such neuropathies are associated with significant physical disabilities, generating high social-economic cost, an important challenge for clinical interventions. Currently, leprosy neuropathies are treated with standard protocols, using either corticoid treatment regimens and/or surgical interventions for nerve decompression. Therefore, LLLT may be a novel auxiliary therapeutic resource in leprosy in order to improve patients' nerve conduction velocity, diminish pain, and minimize physical disabilities, probably reducing the usage period of maximum dose of corticoids, and the number of surgical procedures in the future. Furthermore, this therapeutic approach is also a non-invasive treatment and has a relatively low cost.

Despite the absence of studies on LLLT effects in affected nerves of patients with leprosy, there are some studies showing positive effects in other neuropathies, such as: improvement in clinical and electrophysiological parameters, reduction of pain, improvement of inflammation in nerve entrapment neuropathy, as well as for the promotion of nerve regeneration. Considering that LLLT approach may promote analgesic effects (Chen et al., 2014; Ozkan et al., 2014), improve clinical and electrophysiological parameters (Ozkan et al., 2014; Khamseh et al., 2011), induce anti-inflammatory effects and nerve repair (Chen et al., 2014; Lazovic et al., 2014; Alcântara et al., 2013; Hsieh et al., 2012), and reduce degeneration of the myelin sheat by increasing conduction velocity (Khamseh et al., 2011) in other neuropathologies, we believe that LLLT may also promote the favourable effects in leprosy neuropathy.

This work aims to evaluate the effects of the application of LLLT in the peripheral nerve of leprosy patients. This project was approved N. 989.148/2015 by the Research Ethics Committee of the Federal University of Uberlandia. A randomized, double-blind, placebo-controlled clinical trial will be conducted from January 2017 to December 2019.

The patients will be recruited at the National Reference Centre for Sanitary Dermatology and Leprosy (CREDESH), Federal University of Uberlandia (UFU), State of Minas Gerais, Brazil and then will be informed about the study procedures and will sign the informed consent form. CREDESH is a public health care facility in an endemic region where routine prevention, including intradermal Bacilo Calmette-Guérin (BCG) vaccination, Household Contacts (HHCs) monitoring, early case detection and treatment are available and are under supervision, with multidisciplinary team.

Adult patients (n=92) aged 18-60 years old diagnosed with presence of focal demyelinating neuropathy in compression sites of the ulnar and common peroneal nerves. The patients are selected of household contacts group who became ill during the follow up for 5 to 7 years in the epidemiological surveillance program of the CREDESH/UFU. Clinical dermato-neurological examination, serology anti-PGL-1 are performed annually. When participants present more than one positive result during follow-up, they will undergo in six slit-skin smear sampling for bacilloscopy and quantitative PCR (qPCR) M. leprae DNA with M. leprae-specific repetitive element (RLEP3) detection (lobes of the right and left ears; right and left elbow and right and left knee). Then, the patients are forwarded for dermato-neurological examination, sensitivity and muscle force evaluation (hands, feet and eyes), incapacity degree evaluation, electroneuromyography examination of upper and lower limb. All patients will be treated with multidrug therapy (MDT), according to their operational classification (Paucibacillary - PB and Multibacillary - MB) and their Ridley Jopling classification (tuberculoid and/or borderline tuberculoid (TT), borderline-borderline (BB), borderline lepromatous (BL) and lepromatous (LL)). The patients will be randomized and divided into two groups:

1. Control: patients who will receive application "sham LLLT". The laser will be turned off, but the procedure will be the same as with the LLLT group);
2. LLLT: patients who will receive treatment with LLLT for 12 sessions in alternate days during 4 weeks on nerves:

   1. ulnar nerve: laser probe will be applied around the ulnar nerve at the elbow region, especially in the region of the cubital tunnel at a total of 5 points (3 points above and two points below at medial epicondyle. The distance between of the applications points is 1cm.
   2. common peroneal nerve: will be applied LLLT at 2 points above and 3 points surrounding fibular head. The distance between of the applications points is 1cm. The LLLT will be applied using a diode laser device with parameters: 830 nanometers (nm), 100 milliwatts (mW), 8 Joules (J), 3mW/cm2. Laser probe will be applied directly and perpendicularly in skin contact, the time of irradiation will be 80 seconds per point and treatments will be applied for three times a week for 12 sessions.

ELIGIBILITY:
Inclusion criteria:

* leprosy patients;
* patients who show signs of focal demyelinating neuropathy in compression sites of the ulnar and common peroneal nerves by ENM;
* patients with borderline tuberculoid (BT), borderline-borderline (BB), borderline lepromatous (BL) and lepromatous (LL) leprosy forms;
* patients under multidrug therapy (MDT) and;
* (d) patients who live in Uberlândia (Minas Gerais/Brazil).

Exclusion criteria:

* patient diagnosed with other forms of peripheral neuropathies, diagnosed with diabetes and arterial hypertension;
* patient physically disabled;
* patient with cognitive impairment and;
* who refuse to sign a consent form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Conduction Velocity at 28 days after LLLT. | Patients will be assessed one day before the first day of LLLT application and after 28 days of LLLT application.
  Will be performed on the MEB4200K, the active recording electrode is placed on the center o the muscle belly, and the reference electrode is placed distally, over the muscle tendon. Below is a description of the technique employed in each of these nerves: Ulnar Motor Nerve: Normal values: Amplitude≥ 3.80mv, conduction velocity ≥ 50m/s, distal latency ≤ 3.1 m/s. Delta conduction velocity (difference between the distal segment and the elbow segment)≥10m/s; (b)Common Peroneal Motor Study: Normal values: Amplitude ≥ 2.80 mv, conduction velocity ≥ 40m/s, distal latency(handle)≤ 5.0 msec. Delta conduction velocity (difference between the distal segment and the peroneal head segment)≥10m/s.

SECONDARY OUTCOMES:
Change from Baseline Muscle Strength at 28 days after LLLT. | Patients will be assessed one day before the first day of LLLT application and after 28 days of LLLT application.
  will be assessed muscles innervated by ulnar and common fibular nerves according to the Scale Assessment of Muscular Strength by Kendall et al., 1995. In this scale, there is a score from 0 to 5 that indicates score 5 to complete range of motion against gravity and resistance maxima manual and score 0 without muscle contraction.
Change from Baseline Tactile Sensitivity at 28 days after LLLT. | Patients will be assessed one day before the first day of LLLT application and after 28 days of LLLT application.
  will be used a set of six Semmes-Weinstein monofilaments (Kit prepared by SORRI team, Bauru/SP), to evaluate threshold values for touch. The filament size was marked with the log forces, which are said to represent the threshold values for touch; 0,05 gramas (g) (normal sensation), 0.2g (diminished light touch), 2.0g (diminished protective sensation), 4.00g and 10g(loss of protective sensation of the hands and feet), 300g (feeling of pressure in hand) and black color (no sensation).
  In the tactile sensitivity of ulnar and median nerves , each evaluated point will be received a score from 0 to 5, the final score obtained by summing points : 1,2 and 3 to the median nerve ; 4.5 and 6 for the ulnar nerve , with a maximum score of 15 for each nerve. For the common peroneal nerve will be considered only point 10, with a maximum score of 5. For the tibial nerve will be evaluated 9 points, with a maximum score of 45.
Change from Baseline Pain intensity at 28 days after LLLT. | Patients will be assessed one day before the first day of LLLT application and after 28 days of LLLT application.
  This scale will be used to evaluate the intensity of pain in the innervated region of the ulnar and/or peroneal nerves. There is a score from 0 to 10, 0 indicating no pain and 10 indicating severe pain
Change from Baseline Tissue temperature variations of the body surface at 28 days after LLLT | Patients will be assessed one day before the first day of LLLT application and after 28 days of LLLT application.
  Infrared thermographic consisting of a thermal camera, a computer and a monitor will be used to detect temperature differences after LLLT treatment in leprosy patients. The device calibration is automatic, as recommended by the manufacturer, occurring constantly while connected. A precise thermometer (Minipa®, Brazil) will be used to monitor the room temperature, which will be maintained between 23 and 24 °C. To carry out the acquisition of the thermal images, recommendations of the Brazilian Association of Medical Thermology (ABRATERM) will be followed. The room relative humidity lower than 60% and cutaneous emissivity was set to 0.98. Camera positioned on a tripod 50 cm away from the patient. After we take images, some areas of hands and feet will be chosen on the same anatomical locations for all patientes. The mean ΔTs (temperature differences) for each area will be subsequently calculated (ThermaCAM Researcher Professional, version 2.10, FLIR Systems).
Change from Screening of Activity Limitation and Safety Awareness Scale at 28 days after LLLT. | Patients will be assessed one day before the first day of LLLT application and after 28 days of LLLT application.
  This scale will be used to evaluate of activity limitation and risk awareness. It includes assessment of the eyes, hands, feet (mobility) and self-care. SALSA scores range from 10 to 80, with 10-24 allocated to patients without significant limitations; 25-39 for mild limitations and 40-49; 50- 59 and 60-80 for moderate, severe and very severe limitations, respectively. The risk awareness score ranges from 0 to 11, with higher scores indicating greater awareness of the risks involved in daily life activities.

CONTACTS AND LOCATIONS:
Overall Officials: Isabela M Bernardes Goulart, doctorate, Study Director — Federal University of Uberlandia; Elaine F Sabino, master, Principal Investigator — Federal University of Uberlandia
Locations (1):
- National Reference Center for Sanitary Dermatology and Leprosy, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
This project doesn´t have a plan to make individual participant data available to other researchers. The datas are available only for our researcher group.

REFERENCES:
- [Background] Ozkan FU, Saygi EK, Senol S, Kapci S, Aydeniz B, Aktas I, Gozke E. New treatment alternatives in the ulnar neuropathy at the elbow: ultrasound and low-level laser therapy. Acta Neurol Belg. 2015 Sep;115(3):355-60. doi: 10.1007/s13760-014-0377-9. Epub 2014 Oct 16. PMID 25319131
- [Background] Khamseh ME, Kazemikho N, Aghili R, Forough B, Lajevardi M, Hashem Dabaghian F, Goushegir A, Malek M. Diabetic distal symmetric polyneuropathy: effect of low-intensity laser therapy. Lasers Med Sci. 2011 Nov;26(6):831-5. doi: 10.1007/s10103-011-0977-z. Epub 2011 Aug 19. PMID 21853320